CLINICAL TRIAL: NCT06709300
Title: A Prospective Feasibility Study to Evaluate the Safety and Effectiveness of the ETX-4143 Device in Subjects With Ocular Hypertension
Brief Title: An Observational Study to Evaluate the ETX-4143 Device in Subjects With Ocular Hypertension
Status: Withdrawn | Type: Observational
Why Stopped: Executive decision by the company not to execute the study
Sponsor: EyeCool Therapeutics, Inc. (Industry)
Collaborators: EyeCool Therapeutics, Pty Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: ETX4143-A003
Record Dates: First submitted 2024-10-30; First posted 2024-11-29 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-03

CONDITIONS: Ocular Hypertension
Keywords: Ocular Hypertension; intraocular pressure; Elevated IOP; Eye Diseases; Glaucoma; Raised intraocular pressure
MeSH Terms: conditions — Ocular Hypertension; Eye Diseases; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: Open-label treatment group with the EyeCool ETX-4143 device in eyes with ocular hypertension that meet the inclusion/exclusion criteria

SUMMARY:
This study aims to assess the effectiveness of the EyeCool ETX-4143 device in reducing intraocular pressure (IOP) in eyes with ocular hypertension, regardless of a formal diagnosis of primary open-angle glaucoma. The primary objective is to determine whether the EyeCool device can effectively lower IOP in individuals with elevated eye pressure. Participants currently using intraocular pressure-lowering medications but still experiencing elevated IOP may also be eligible to participate.

DETAILED DESCRIPTION:
This is a prospective feasibility study designed to evaluate the safety and effectiveness of the EyeCool ETX-4143 device in lowering intraocular pressure (IOP) in eyes with ocular hypertension.

Elevated IOP can negatively affect the optic nerve, often resulting from various clinical conditions. The progression of IOP elevation is typically gradual and painless, which may lead to it going unnoticed by the patient. If left untreated, significantly elevated IOP can cause permanent visual field reduction and vision loss.

Ocular hypertension may occur with or without a formal diagnosis of primary open-angle glaucoma. Additionally, individuals with ocular hypertension may or may not be on ocular hypotensive medications to manage their condition.

This exploratory study aims to determine whether treatment with the EyeCool device results in a safe and effective reduction in IOP. Up to 30 eyes with ocular hypertension will be enrolled and followed for 12 weeks after treatment.

If both eyes meet the inclusion and exclusion criteria, only the eye with the higher IOP will be treated. Participants will not be required to discontinue or modify their use of IOP-lowering medications during the study.

Study findings are expected to inform the design of future clinical trials assessing the ETX-4143 device for the treatment of elevated IOP.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients age ≥40 years of age of any gender
2. Has been diagnosed with elevated IOP (all readings should be taken within the same 4hr daytime window) with a reading of > 21mm Hg in the eye to be studied.
3. Is either not being treated for elevated IOP or is using ocular hypotensive medication to control IOP.
4. Have an open angle of the anterior chamber with evidence of trabecular meshwork visible on gonioscopy
5. Willing to forgo participation in any other clinical study for the duration of this study
6. Demonstrate sufficient cognitive awareness to comply with the examination process
7. Willing and able to comply with schedule for follow-up visits
8. Willing to participate in the study as evidenced by signing of an informed consent document

   Exclusion Criteria:
9. Women who are pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study time period, including the follow-up period
10. Known allergy or hypersensitivity to copper, aluminum, or silicone
11. Have previously undergone penetrating intraocular glaucoma surgeries (e.g., glaucoma filtering surgery, trabeculectomy, or tube bypass) in any quadrant of the study eye
12. Have undergone laser trabeculoplasty (ALT, MLT, or SLT, or cilio-ablative therapy such as cyclophotocoagulation (CPC)) within 90 days prior to starting the study
13. Any active ocular infection (bacterial, viral, or fungal), or active ocular inflammation at the time of the Screening Visit (note- potential subjects can return for rescreening at a later date after the infection or inflammation has resolved.)
14. History of corneal transplant (penetrating keratoplasy or endothelial keratoplasty), significant corneal endothelial disease, keratoconus, corneal thinning, or other corneal ectasias
15. A history of herpes keratitis, non-healing corneal epithelial defects, or neurotrophic keratopathy due to corneal herpetic disease, stem cell deficiency, diabetic keratopathy, severe lagophthalmos, topical anesthetic abuse, or any other cause
16. Any history of significant conjunctival surgery within the prior 90 days such as pterygium removal, or any presence of any subconjunctival implant (scleral buckle surgery).
17. Planned eye surgery or other ophthalmic procedures within 90 days following treatment.
18. Participation in any clinical study of an investigational product within 30 days prior to enrollment
19. Any history of serious, poorly controlled systemic or ophthalmic condition or circumstances, including those identified in the screening visit which, in the opinion of the Investigator, could compromise the subject's ability to comply with the protocol or that could compromise the subject's safety or the interpretation of the clinical trial results.
20. Neuropsychiatric disorder (e.g. psychosis, schizophrenia, mania, depression) or major psychiatric illness that has required hospitalization within the last 6 months prior to screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals that have been diagnosed with hypertension and are seen in the general patient population of an ophthalmic primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Individual percent reduction in IOP | From treatment to the end of twelve weeks
  Individual percent reduction in intraocular pressure at each post-treatment exam compared to baseline while maintaining the same concomitant ocular hypotensive medication regimen, if any.
Mean reduction in intraocular pressure | From treatment to the end of twelve weeks
  Mean reduction in IOP at each post-treatment exam compared to baseline while maintaining the same concomitant ocular hypotensive medication regime, if any.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick R Casey, OD, Study Chair — EyeCool Therapeutics, Inc.
Locations (1):
- Ophthalmic Trials Australia, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No